CLINICAL TRIAL: NCT01562210
Title: Olaparib Dose Escalating Trial in Patients Treated With Radiotherapy With or Without Daily Dose Cisplatin for Locally Advanced Non-small Cell Lung Carcinoma
Brief Title: Olaparib Dose Escalating Trial + Concurrent RT With or Without Cisplatin in Locally Advanced NSCLC
Acronym: olaparib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL35195.031.11; N11ORL (Registry Identifier: PTC)
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: NSCLC
Keywords: NSCLC; Olaparib; CCRT
MeSH Terms: interventions — olaparib; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olaparib, radiation +/- Cisplatin (Experimental): Olaparib and radiotherapy with or without Cisplatin
  Interventions: Drug: Olaparib; Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Olaparib — Olaparib will be given orally BID for 36 days, administrated with a 12 hour interval. Olaparib will start 2 days before RT and will continue for 2 days after the last RT fraction. Olaparib is also given during the non-radiotherapy days but no maintenance treatment is given after radiotherapy is finished.
  The first cohort will receive Olaparib with a dose of 25mg BID combined with Cisplatin and RT. Thereafter in both with and without cisplatin arms dose escalation will follow to 50mg, 100mg, 200mg, 300mg and 400mg BID.
  Other Names: AZD2281
Drug: Cisplatin — 6 mg/m2 (5 days/week), 1-1.5 hr before the irradiation (week 1 to 5), given as a 5-minutes intravenous infusion.
  Other Names: L01XA03
Radiation: Radiation — A total dose of 66 Gy will be given in 24 fractions from week 1 to 5, excluding the weekends.

SUMMARY:
Phase I dose escalating trial. Primary objective of this study is to define the maximal tolerated dose (MTD)of Olaparib in combination with high dose radiotherapy with or without daily dose Cisplatin in locally advanced NSCLC. Secondary objectives include to define safety profile, determine PK/Pd variables and document preliminary evidence of objective tumor response.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy (CCRT) is the treatment of choice for patients with locally advanced NSCLC. The cure rates however need to be improved. The main mechanism by which both radiation and Cisplatin kill tumor cells is by an accumulation of un- or misrepaired DNA damage.PARP inhibitors increase radiation and chemotherapy (Cisplatin) response in preclinical studies including lung cancer models.

This open label dose escalating trial consists of a screening phase, a treatment phase and a follow up phase.

The screening phase: patients who can tolerate concurrent cisplatin will receive Olaparib, RT and Cisplatin. Patients who can not tolerate concurrent cisplatin will receive Olaparib and RT with or without prior sequential chemotherapy.

The treatment phase:dose escalation of Olaparib will be performed in cohorts of 3 subjects. The decision to escalate to the next dose level will be based on the occurrence of DLTs during the DLT evaluation period (i.e. 3 months following the last day of irradiation) and will be made after all patients within the cohort have completed their third month of follow up.

Active follow-up phase: frequent follow up will take place during the first 3 months (acute toxicity). Thereafter patients will be monitored for late toxicity and for disease activity 3-monthly throughout the first year and thereafter 6-monthly until 5 years, when patients are deemed to be cured and follow up is no longer warranted.

Olaparib will be given orally BID for 36 consecutive days, administrated with a 12 hour interval. Olaparib will start 2 days before start of RT and will continue for 2 days after the last RT fraction. Olaparib is also given during the non-radiotherapy days but no maintenance treatment is given after radiotherapy is finished.

Radiotherapy (for all patients): a total dose of 66Gy will be given in 24 fractions from week 1 to 5.

Cisplatin (concurrent chemoradiotherapy): daily dose Cisplatin 6mg/m2 (5 days/week), 1-1.5 hr before the irradiation (week 1 to 5), given as a 5-minutes intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Histologically or cytologically confirmed diagnosis of NSCLC
* Stage II/III non-operable disease, without malignant pleural effusion
* Presence of at least one measurable target lesion
* Acceptable pulmonary function as defined by a Fev1 of ≥30% and a DLCO of ≥ 40% of predicted,
* NYHA I-II functional status
* Expected risk of radiation-induced pulmonary toxicity is modest: MLD ≤ 20 and maximum cord dose 50 Gy
* WHO performance 0-1
* Life expectancy of at least 6 months
* Adequate hematological, renal and hepatic functions

  * Hemoglobin ≥ 5.5 mmol/l
  * Leucocytes > 3.0 x 109/l
  * Absolute neutrophil count > 1.5x109/l
  * Platelet count > 100 x 109/l
  * Total bilirubin < 1.5 x UNL
  * ASAT/ALAT < 2.5 x UNL
  * Alkaline phosphatase < 5 x UNL
  * Creatinine < 130 mmol/l or creatinine clearance > 50 ml/min; measured or calculated
  * Urine dipstick for proteinuria < 2+. If urine dipstick is ≥ 2, 24 hour urine must demonstrate < 500 mg of protein in 24 hours
* No pre-existing sensory neurotoxicity grade ≥ 1 (CTCAE)
* Patients of reproductive potential must agree to practice two effective medically approved contraceptive method during the trial and 3 months afterwards
* Signed written informed consent.

Exclusion Criteria:

* Concurrent active malignancy other than localized, non-melanoma skin cancer or carcinoma-in-situ of the cervix (unless definitive treatment was completed 5 years or more before study entry and the patient has remained disease free)
* Anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the 3 weeks prior to start of therapy (or a longer period depending on the defined characteristics of the agents used e.g. 6 weeks for mitomycin or nitrosourea). Patients may continue the use of LHRH agonists for cancer; bisphosphonates for bone disease and corticosteroids.
* Patients, selected for sequential chemoradiotherapy, are excluded if no disease control (all responses except progression) is obtained after induction chemotherapy.
* Prior:

  * Ipsilateral radiotherapy to the chest;
  * Chemotherapy for other indications than NSCLC within the last 5 years
* History of interstitial pneumonitis (to include diffuse alveolar damage, non-malignant causes of pneumonitis, ARDS, alveolitis, cryptogenic organising pneumonia, obliterative bronchiolitis, non-malignant causes of pulmonary fibrosis, eligibility based on the judgement of the primary investigator), active infection on day of enrolment
* Significant cardiovascular disease as defined by:

  * History of congestive heart failure requiring therapy;
  * History of unstable angina pectoris or myocardial infarction up to 6 months prior to trial entry;
  * Presence of severe valvular heart disease;
  * Presence of a ventricular arrhythmia requiring treatment;
  * Uncontrolled hypertension
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed with the patient before registration in the trial.
* Participation in other trial with investigational drug or treatment modality
* Co-existing serious active infection requiring parenteral antibiotics
* Patients with hepatic disease e.g. patients with known serologically positive Hepatitis B or Hepatitis C as they may be more at risk of toxicity from Olaparib
* Immunocompromised patients e.g. human immunodeficiency virus (HIV)
* Myelodysplastic syndrome/acute myeloid leukaemia or features suggestive of MDS/AML on peripheral blood smear.
* Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study
* Gastrointestinal disorders that may interfere with absorption of the study drug or patients who are not able to take oral medication
* Concomitant medications:

  * Any previous treatment with a PARP inhibitor, including Olaparib
  * Patients receiving the following classes of inhibitors of CYP3A4 (see Section 7.4 for guidelines and wash out periods)

    * Azole antifungals
    * Macrolide antibiotics
    * Protease inhibitors
* Persistent grade 2 or greater toxicities, from any cause
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-04; Primary Completion 2019-05 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
The incidence of dose limiting toxicities (DLTs) | from start until 3 months after the last RT day
  The incidence of dose limiting toxicities occuring during the DLT evaluation period (from start of study treatment until 3 months after the last radiation day). This endpoint will be used to determine the maximal tolerated dose of Olaparib in combination with radiotherapy with and without low dose Cisplatin.

SECONDARY OUTCOMES:
Additional safety variables | until 5 years after treatment
  (S)AE's, laboratory parameters, vital signs, lung function, long term toxicity: defined as grade ≥ 2 toxicity (with a special attention for pulmonary and esophageal toxicity) that is possibly, probably or definitely related to study treatment, occurring or persisting from 3 months after the last irradiation day until 5 years after treatment.
Objective tumor response | until 5 years after treatment
Locoregional control rate (LRCR) | at one year
Progression free survival | until 5 years after treatment
Pharmacokinetic variables | week -1 (baseline) until week 11
  AUC, Cmax, Cmin
Pharmacodynamic variables | week -1 (baseline) until week 8
  PARP inhibition, γH2AXfoci formation
Surrogate biomarkers for antitumor response | until 5 years after treatment
  metabolic response determined by FDG-PET/CT-imaging, change in circulating tumor cells, molecular/biological parameters (tumor markers)

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Verheij, MD, PhD, Principal Investigator — Antoni van Leeuwenhoekziekenhuis (NKI-AVL); Michel M. van den Heuvel, MD, PhD, Principal Investigator — Antoni van Leeuwenhoekziekenhuis (NKI-AVL)
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Ziekenhuis (NKI-AVL), Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van Werkhoven E, Hinsley S, Frangou E, Holmes J, de Haan R, Hawkins M, Brown S, Love SB. Practicalities in running early-phase trials using the time-to-event continual reassessment method (TiTE-CRM) for interventions with long toxicity periods using two radiotherapy oncology trials as examples. BMC Med Res Methodol. 2020 Jun 22;20(1):162. doi: 10.1186/s12874-020-01012-z. PMID 32571298
- [Derived] de Haan R, van Werkhoven E, van den Heuvel MM, Peulen HMU, Sonke GS, Elkhuizen P, van den Brekel MWM, Tesselaar MET, Vens C, Schellens JHM, van Triest B, Verheij M. Study protocols of three parallel phase 1 trials combining radical radiotherapy with the PARP inhibitor olaparib. BMC Cancer. 2019 Sep 10;19(1):901. doi: 10.1186/s12885-019-6121-3. PMID 31500595